CLINICAL TRIAL: NCT06132659
Title: Neurofeedback Enhanced Cognitive Reappraisal Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Stefanie Russman Block, Clinical Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00209563
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Social Anxiety Disorder; Panic Disorder; Generalized Anxiety Disorder
Keywords: functional magnetic resonance imaging
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Masking Description: (Veritable-NF (MPC) and Sham-NF only): All staff present during the MRI session, as well as the participant, will be blinded to group assignment. A designated member of the study team will remain unblinded during the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Veritable-NF (MPC) (Experimental)
  Interventions: Other: Functional magnetic resonance imaging (fMRI) with Veritable-NF
- Sham-NF (Active Comparator)
  Interventions: Other: fMRI with Sham-NF
- Veritable-NF (PFC) (Active Comparator)
  Interventions: Other: Functional magnetic resonance imaging (fMRI) with Veritable-NF

INTERVENTIONS:
Other: Functional magnetic resonance imaging (fMRI) with Veritable-NF — Participants will have 4 visits (some can be done virtually). The baseline visit will include an interview and questionnaires. Eligible participants will have a practice session at visit 2, and may do a mock scanner if the visit is in person. Visit 3 will take place within 5 days of the practice session and participants will be asked to complete questionnaires and have an fMRI with the real neurofeedback. Visit 4 will take place one month after visit 3 and will include a follow-up interview with a trainer assessor as well as questionnaires. Additionally, 2 weeks after visit 3 participants will also complete some questionnaires online.
  Arms: Veritable-NF (MPC); Veritable-NF (PFC)
Other: fMRI with Sham-NF — Participants will have 4 visits (some can be done virtually). The baseline visit will include an interview and questionnaires. Eligible participants will have a practice session at visit 2, and may do a mock scanner if the visit is in person. Visit 3 will take place within 5 days of the practice session and participants will be asked to complete questionnaires and have an fMRI with feedback that looks similar to real neurofeedback, but is computer generated. Visit 4 will take place 2 weeks after visit 3 and participants will complete more questionnaires.
  Arms: Sham-NF

SUMMARY:
This study seeks to understand emotion regulation in those with anxiety using real-time functional magnetic resonance imaging neurofeedback, a tool that allows individuals to control brain activity. The goal of this project is to understand how receiving feedback about one's own brain activity relates to emotion regulation ability. This work will help the study team understand the brain areas involved in emotion regulation and could lay the groundwork to test if psychotherapy outcomes can be enhanced using neurofeedback.

The study hypotheses include:

* Participants receiving veritable-Neurofeedback (NF) will show a greater activation increase in the prefrontal cortex (PFC) compared to sham-NF
* Participants receiving veritable-NF will show greater cognitive reappraisal (CR) ability compared to those receiving sham-NF
* Prefrontal cortex activation will positively correlate with CR ability

DETAILED DESCRIPTION:
Due to an unforeseen error in our online neurofeedback script, in which the location of the brain region being targeted was not properly read by the script, participants in the veritable-NF group received feedback to the medial parietal cortex (MPC) instead of the PFC. A third, unrandomized arm has been added to this registration to enroll an additional subset of participants who are indeed receiving feedback to the PFC. The pre-existing veritable-NF arm has been relabeled to reflect which region of the brain was actually targeted. Additionally, the masking description has been reset to "None".

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis (primary source of distress and/or interference) of generalized anxiety disorder, social anxiety disorder, panic disorder or illness anxiety disorder based on structured interview. Comorbid phobic disorders allowed, but these cannot be the primary source of interference or distress due to the lowered chances of encountering anxiety-provoking stimuli during the study period
* Score of 2 or more on at least 1 question from the GAD/CROSS-AD composite
* Medically and physically able to consent
* Not regularly taking any medication, prescription or non-prescription, with psychotropic effects other than:

  1. Buspirone, or antidepressant (e.g., selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI)) with stable dosage for past 4 weeks
  2. Hormonal contraceptives of any type for any duration
* For females, not currently pregnant or actively trying to become pregnant
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition (per protocol)
* Size compatible with scanner gantry (per protocol)

Exclusion Criteria:

* Current diagnosis of Obsessive Compulsive Disorder, Posttraumatic Stress Disorder, or Bipolar Disorder
* Current substance abuse or dependence (past 6 months)
* Active suicidality with plan or intent
* Current psychosis
* History of serious neurological illness or current medical condition that could compromise brain function, such as liver failure
* History of closed head injury, e.g., loss of consciousness greater (>) approximately (~) 5 minutes, hospitalization, neurological sequela

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Russman Block, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Veritable-NF (MPC) | Sham-NF | Veritable-NF (PFC)
Started | 7 | 6 | 8
Completed | 7 | 5 | 8
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veritable-NF (MPC) | Sham-NF | Veritable-NF (PFC) | Total
Number analyzed (Participants) | 7 | 6 | 8 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 8 | 21
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (11.6) | 30.3 (11.9) | 28.3 (8.9) | 28.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 15
  Male | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 7 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 8 | 21
Hamilton Anxiety Rating Scale [Mean (Standard Deviation); unit: score on a scale] — Total score is reported. Scores range from 0-56 and higher scores represent greater anxiety symptoms severity.
  score on a scale | 13.29 (8.83) | 14.50 (9.33) | 16.88 (9.06) | 15.00 (8.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in Prefrontal Cortex (PFC) Activity (Baseline to Transfer Run) From the Reappraise > Look Contrast on the Emotion Regulation Task (ERT)
Description: The PFC was defined in MNI space using significant group level activation in the posterior medical frontal cortex from the reappraise>look contrast from earlier pilot subjects. Percent signal change in this region was extracted for all participants. Change in PFC activity was calculated as the linear slope of change across all 5 runs of the task. To this end, a linear regression was conducted for each participant separately with "run" as the independent variable and "PFC percent signal change" as the dependent variable to calculate change in percent signal change over time. These slopes were then averaged for each group .
Time Frame: Approximately 60 minutes
Population: 1 participant in the sham group had too much motion during the neurofeedback runs of the scans to be included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent signal change per run
Arm/Group | Veritable-NF (MPC) | Sham-NF | Veritable-NF (PFC)
Number analyzed (Participants) | 7 | 5 | 8
Percent signal change per run | 0.042 (0.077) | 0.019 (0.056) | 0.007 (0.075)

2. Primary Outcome: Difference in Negative Affect Ratings of Images From International Affective Picture System (IAPS)
Description: The Self-Assessment Manikin (SAM) is a pictorial assessment technique in which a changing manikin figure depicts values along the primary dimension of affective valence (positive/negative). Users may indicate emotional reactions along a scale from 1-9, with higher numbers indicating greater negative affect. After the scan, participants will rate each image they saw along this scale. Differences in SAM ratings from look to reappraise trials (e.g., average reappraise score minus average look score) will be evaluated and compared between sham-NF and veritable-NF groups. Higher difference score indicates that images viewed during reappraisal are seen as more positive than those viewed during the look condition.
Time Frame: Within 10 minutes of exiting the scanner
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veritable-NF (MPC) | Sham-NF | Veritable-NF (PFC)
Number analyzed (Participants) | 7 | 6 | 8
score on a scale | 0.57 (0.73) | 0.29 (0.26) | 0.03 (0.35)

3. Secondary Outcome: Change in Amygdala-PFC Functional Connectivity (Baseline to Transfer) From Reappraise > Look Contrast
Description: To examine amygdala connectivity, the study team will use a psychophysiological interaction analysis. Deconvolved time series from anatomical left and right amygdala seeds for each participant will be multiplied by a vector for the reappraise > look contrast at each run (baseline, neurofeedback (NF1, NF2, NF3), transfer). Regressors for the seed time series, the original condition and the interaction term will be convolved with the canonical hemodynamic response function. Change in connectivity from pre-to-post training will be calculated by subtracting the baseline-run contrast map from the transfer-run contrast map. Resulting contrast maps will be entered into second-level random effects analyses in the software SPM, where voxels in the PFC will be examined at p<0.05 FWE-corrected threshold.
Time Frame: Each run is approximately 9 minutes long. Run 5 starts approximately 30 minutes after the completion of run 1.
Population: as for outcome 1
Measure: Number; unit: Number of significant voxels in the PFC
Arm/Group | Veritable-NF (MPC) | Sham-NF | Veritable-NF (PFC)
Number analyzed (Participants) | 7 | 5 | 8
Number of significant voxels in the PFC | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Veritable-NF (MPC) | Sham-NF | Veritable-NF (PFC)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 1/6 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veritable-NF (MPC) (N=7) | Sham-NF (N=6) | Veritable-NF (PFC) (N=8)
Foot abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Participant presented to the emergency room for foot abscess after consent, but prior to the MRI portion of the study. This adverse event was unrelated to the study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT06132659/Prot_SAP_000.pdf